CLINICAL TRIAL: NCT02763215
Title: Multi-Center Study for the Assessment of Copper Parameters in Wilson Disease Subjects on Standard of Care Treatment
Brief Title: The Assessment of Copper Parameters in Wilson Disease Participants on Standard of Care Treatment
Status: Completed | Type: Observational
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: WTX101-203
Record Dates: First submitted 2016-05-03; First posted 2016-05-05 (Estimated); Results first posted 2020-10-26 (Actual); Last update posted 2020-12-01 (Actual); Status verified 2020-11

CONDITIONS: Wilson Disease
MeSH Terms: conditions — Hepatolenticular Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Total
  Interventions: Drug: Standard of Care Medications

INTERVENTIONS:
Drug: Standard of Care Medications — Standard of care medications could include penicillamine, trientine, zinc, or a combination of a copper chelator and zinc.

SUMMARY:
This was a 24-month study to assess copper parameters in participants with Wilson disease (WD) treated with standard of care (SoC) medications.

After providing informed consent, participants meeting all inclusion and no exclusion criteria were enrolled into the study as outpatients. The participants' routine clinic visits were scheduled according to the standard clinical practice at the study center and at the discretion of the treating physician at approximate 6-month intervals.

At the time of enrollment, participants were receiving SoC medications for the treatment of WD, which could include penicillamine, trientine, zinc, or a combination of a copper chelator and zinc. If treatment was interrupted or stopped during the course of the study, participants continued in the study and biological samples and clinical data were continued to be collected for the full 24-month study period. Dosing with SoC agents was individualized and managed by the treating physician at the study center according to standard clinical practice at the site.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to give informed consent for participation in the study.
* Male or female participants, aged 18 years or older as of signing the informed consent form.
* Receiving SoC medications (penicillamine, trientine, zinc, or copper chelators with zinc) for the treatment of WD at the time of enrollment and for no more than 60 months prior to enrollment.
* Able to understand and willing to comply with study procedures and requirements, as judged by the Investigator.
* Established diagnosis of WD.
* Adequate venous access to allow for collection of blood samples.

Exclusion Criteria:

* Major systemic disease or other illness that would, in the opinion of the Investigator, compromise participant safety or interfere with the collection or interpretation of study results.
* In the opinion of the Investigator, the participant was likely to be non-compliant or uncooperative during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Wilson disease participants receiving SoC medications for the treatment of WD. Standard of care medications could include penicillamine, trientine, zinc, or a combination of a copper chelator and zinc.
Sampling Method: Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2016-05-19 (Actual); Primary Completion 2019-01-21 (Actual); Study Completion 2019-01-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexion Pharmaceuticals, Inc., Study Director — Alexion Pharmaceuticals, Inc.
Locations (10):
- United States (5):
  - Clinical Trial Site, New Haven, Connecticut
  - Clinical Trial Site, Chicago, Illinois
  - Clinical Trial Site, Ann Arbor, Michigan
  - Clinical Trial Site, Nashville, Tennessee
  - Clinical Trial Site, Seattle, Washington
- Clinical Trial Site, Vienna, Austria
- Clinical Trial Site, Heidelberg, Germany
- Clinical Trial Site, Warsaw, Poland
- United Kingdom (2):
  - Clinical Trial Site, Birmingham
  - Clinical Trial Site, Guildford

RESULTS

PARTICIPANT FLOW:
Groups:
- Total: Participants in this study were not treated with any investigational products, but with standard of care (SoC) medications, which could include penicillamine, trientine, zinc, or a combination of a copper chelator and zinc.
Period: Overall Study
Arm/Group | Total
Started | 64
Completed | 57
Not Completed | 7
Not completed — Participants withdrew from study | 3
Not completed — Missed visit | 1
Not completed — Visit outside visit-window | 1
Not completed — Death | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Population: Full Analysis Set: Participants enrolled in the study. To be eligibly enrolled, participants must have been receiving the SoC medications (penicillamine, trientine, zinc, or copper chelators with zinc) for the treatment of WD at the time of enrollment and for no more than 60 months prior to enrollment.
Groups:
- Total: Participants in this study were not treated with any investigational products, but with SoC medications, which could include penicillamine, trientine, zinc, or a combination of a copper chelator and zinc.
Arm/Group | Total
Number analyzed (Participants) | 64
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.0 (11.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36
  Male | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 62
  Unknown or Not Reported | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian | 2
  Race: Black or African American | 1
  Race: White | 57
  Race: Other | 4

OUTCOME MEASURES:

1. Primary Outcome: Percentage Of Participants Who Achieved Or Maintained Normalized Concentrations Of Non-ceruloplasmin-bound Copper (NCC) Or Reached A Reduction Of ≥ 25% In NCC During 6 Months Of Treatment
Description: To achieve a normalized NCC concentration, participants must have had 2 consecutive measures within (or below) the normal concentration range (0.8 to 2.3 micromolar [μM]). Two consecutive measurements required that the measurements occurred on separate dates and were assigned to 2 different visits. Non-ceruloplasmin-bound copper was calculated by subtracting the amount of copper bound to the ceruloplasmin from the total plasma copper concentration.
Time Frame: Baseline through Month 6
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Total
Number analyzed (Participants) | 64
Percentage of participants | 51.6 [51.2 to 78.8]

2. Secondary Outcome: Percentage Of Participants Who Achieved Or Maintained Normalized Concentrations Of NCC Or Reached A Reduction Of ≥ 25% In NCC Through Last Assessment
Description: To achieve a normalized NCC concentration, participants must have 2 consecutive measures within (or below) the normal range (0.8 to 2.3 μM). Two consecutive measurements required that the measurements occurred on separate dates and were assigned to 2 different visits. Non-ceruloplasmin-bound copper was calculated by subtracting the amount of copper bound to the ceruloplasmin from the total plasma copper concentration. Last Assessment was the last available post-baseline result for each participant (ranging from 1 to 24 months).
Time Frame: Baseline through Last Assessment (ranging from 1 to 24 months)
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Total
Number analyzed (Participants) | 64
Percentage of participants | 62.5 [59.0 to 83.9]

3. Secondary Outcome: Change From Baseline In NCC Concentrations At Month 6, Month 24, And Last Assessment
Description: Evaluation of NCC concentrations over time are reported as micromoles/liter (μmol/L). Last Assessment was the last available post-baseline result for each participant (ranging from 1 to 24 months).
Time Frame: Baseline through Last Assessment (ranging from 1 to 24 months)
Population: Full Analysis Set: Enrolled participants. To be eligibly enrolled, participants must have been receiving the SoC medications (penicillamine, trientine, zinc, or copper chelators with zinc) for the treatment of WD at the time of enrollment and for no more than 60 months prior to enrollment. The number of participants analyzed per row represents number of overall participants continuing in the study at each timepoint with non-missing and non-negative baseline and post-baseline values for NCC.
Measure: Mean (Standard Deviation); unit: μmol/L
Arm/Group | Total
Number analyzed (Participants) | 64
μmol/L
  Month 6: number analyzed (Participants) | 34
  Month 6 | -0.60 (1.441)
  Month 24: number analyzed (Participants) | 29
  Month 24 | -1.24 (1.905)
  Last Assessment: number analyzed (Participants) | 44
  Last Assessment | -0.94 (1.811)

4. Secondary Outcome: Time To Normalization Of NCC If Above The Reference Range At The Time Of Enrollment
Description: The time to normalization of NCC was measured by Kaplan-Meier analysis.
Time Frame: Baseline, up to 24 months
Population: Full Analysis Set with an elevated NCC at Baseline.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Total
Number analyzed (Participants) | 12
Days | 139.5 [62.0 to 545.0]

5. Secondary Outcome: Change From Baseline In Exchangeable Copper At Month 6, Month 24, And Last Assessment
Description: The change in exchangeable copper was evaluated over time and is reported as nanograms/milliliter (ng/mL). Last Assessment was the last available post-baseline result for each participant (ranging from 1 to 24 months).
Time Frame: Baseline through Last Assessment (ranging from 1 to 24 months)
Population: Full Analysis Set: Enrolled participants. To be eligibly enrolled, participants must have been receiving the SoC medications (penicillamine, trientine, zinc, or copper chelators with zinc) for the treatment of WD at the time of enrollment and for no more than 60 months prior to enrollment. The number of participants analyzed per row represents number of overall participants continuing in the study at each timepoint with non-missing baseline and post-baseline values for each outcome measure.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Total
Number analyzed (Participants) | 64
ng/mL
  Month 6: number analyzed (Participants) | 58
  Month 6 | -7.9 (26.02)
  Month 24: number analyzed (Participants) | 53
  Month 24 | -9.5 (27.61)
  Last Assessment: number analyzed (Participants) | 61
  Last Assessment | -8.3 (27.25)

6. Secondary Outcome: Change From Baseline In Copper Plasma Ultrafiltrate At Month 6, Month 24, And Last Assessment
Description: Change in copper plasma ultrafiltrate was measured over time and is reported as ng/mL. Last Assessment was the last available post-baseline result for each participant (ranging from 1 to 24 months).
Time Frame: Baseline through Last Assessment (ranging from 1 to 24 months)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Total
Number analyzed (Participants) | 64
ng/mL
  Month 6: number analyzed (Participants) | 59
  Month 6 | -3.96 (13.082)
  Month 24: number analyzed (Participants) | 53
  Month 24 | 0.00 (30.295)
  Last Assessment: number analyzed (Participants) | 62
  Last Assessment | -0.68 (28.470)

7. Secondary Outcome: Change From Baseline In Plasma Total Copper Used To Calculate NCC At Month 6, Month 24, And Last Assessment
Description: Plasma total copper was measured over time and is reported as ng/mL. Last Assessment was the last available post-baseline result for each participant (ranging from 1 to 24 months).
Time Frame: Baseline through Last Assessment (ranging from 1 to 24 months)
Population: as for outcome 5
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Total
Number analyzed (Participants) | 64
ng/mL
  Month 6: number analyzed (Participants) | 57
  Month 6 | 0.0 [-48.0 to 33.0]
  Month 24: number analyzed (Participants) | 53
  Month 24 | 0.0 [-76.0 to 19.0]
  Last Assessment: number analyzed (Participants) | 61
  Last Assessment | 0.0 [-76.0 to 36.0]

8. Secondary Outcome: Change From Baseline In Serum Total Ceruloplasmin (Nephelometry) Used To Calculate NCC At Month 6, Month 24, And Last Assessment
Description: The total serum (nephelometry) was measured over time and is reported as milligrams (mg)/L. Last Assessment was the last available post-baseline result for each participant (ranging from 1 to 24 months).
Time Frame: Baseline through Last Assessment (ranging from 1 to 24 months)
Population: as for outcome 5
Measure: Median (Inter-Quartile Range); unit: mg/L
Arm/Group | Total
Number analyzed (Participants) | 64
mg/L
  Month 6: number analyzed (Participants) | 62
  Month 6 | 0.0 [-4.0 to 14.0]
  Month 24: number analyzed (Participants) | 56
  Month 24 | 0.0 [-4.5 to 20.5]
  Last Assessment | 0.0 [-4.5 to 20.0]

9. Secondary Outcome: Change From Baseline In 24-Hour Urinary Copper At Month 6, Month 24, And Last Assessment
Description: Evaluation of 24-hour urinary copper over time is reported as micrograms (μg)/day. Last Assessment was the last available post-baseline result for each participant (ranging from 1 to 24 months).
Time Frame: Baseline through Last Assessment (ranging from 1 to 24 months)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: μg/day
Arm/Group | Total
Number analyzed (Participants) | 64
μg/day
  Month 6: number analyzed (Participants) | 50
  Month 6 | -64.7 (353.63)
  Month 24: number analyzed (Participants) | 45
  Month 24 | -113.4 (295.76)
  Last Assessment: number analyzed (Participants) | 55
  Last Assessment | -100.2 (333.70)

10. Secondary Outcome: Change From Baseline In Plasma Total Molybdenum At Month 6 And Month 24
Description: The plasma total molybdenum was measured over time and is reported in ng/mL.
Time Frame: Baseline, Month 6, Month 24
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Total
Number analyzed (Participants) | 64
ng/mL
  Month 6: number analyzed (Participants) | 57
  Month 6 | -4.9 (25.60)
  Month 24: number analyzed (Participants) | 53
  Month 24 | -5.2 (26.53)

11. Secondary Outcome: Change From Baseline In Molybdenum Plasma Ultrafiltrate At Month 6 And Month 24
Description: The molybdenum plasma ultrafiltrate was measured over time and is reported as ng/mL.
Time Frame: Baseline, Month 6, Month 24
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Total
Number analyzed (Participants) | 64
ng/mL
  Month 6: number analyzed (Participants) | 59
  Month 6 | -2.50 (10.963)
  Month 24: number analyzed (Participants) | 53
  Month 24 | -2.89 (11.163)

12. Secondary Outcome: Change From Baseline In 24-Hour Urinary Molybdenum At Month 6 And Month 24
Description: Evaluation of 24-hour urinary molybdenum over time is reported as μg/day.
Time Frame: Baseline, Month 6, Month 24
Population: as for outcome 5
Measure: Median (Inter-Quartile Range); unit: μg/day
Arm/Group | Total
Number analyzed (Participants) | 64
μg/day
  Month 6: number analyzed (Participants) | 48
  Month 6 | 2.5 [-11.5 to 25.0]
  Month 24: number analyzed (Participants) | 44
  Month 24 | 2.0 [-18.5 to 21.0]

13. Secondary Outcome: Change From Baseline In Hepatic Laboratory Measures For Alanine Aminotransferase (ALT) At Month 6, Month 24, And Last Assessment
Description: The ALT levels were measured over time and are reported as units (U)/L. Last Assessment was the last available post-baseline result for each participant (ranging from 1 to 24 months).
Time Frame: Baseline through Last Assessment (ranging from 1 to 24 months)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Total
Number analyzed (Participants) | 64
U/L
  Month 6: number analyzed (Participants) | 61
  Month 6 | 0.8 (29.53)
  Month 24: number analyzed (Participants) | 56
  Month 24 | -1.6 (28.09)
  Last Assessment | -1.5 (28.55)

14. Secondary Outcome: Change From Baseline In Hepatic Laboratory Measures For Aspartate Aminotransferase (AST) At Month 6, Month 24, And Last Assessment
Description: The AST levels were measured over time and are reported as U/L. Last Assessment was the last available post-baseline result for each participant (ranging from 1 to 24 months).
Time Frame: Baseline through Last Assessment (ranging from 1 to 24 months)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Total
Number analyzed (Participants) | 64
U/L
  Month 6: number analyzed (Participants) | 61
  Month 6 | 0.3 (12.69)
  Month 24: number analyzed (Participants) | 56
  Month 24 | -0.7 (11.86)
  Last Assessment | -0.6 (12.54)

15. Secondary Outcome: Change From Baseline In Hepatic Laboratory Measures For Bilirubin At Month 6, Month 24, And Last Assessment
Description: Bilirubin was measured over time and is reported as μmol/L. Last Assessment was the last available post-baseline result for each participant (ranging from 1 to 24 months).
Time Frame: Baseline through Last Assessment (ranging from 1 to 24 months)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: μmol/L
Arm/Group | Total
Number analyzed (Participants) | 64
μmol/L
  Month 6: number analyzed (Participants) | 61
  Month 6 | 0.2 (6.10)
  Month 24: number analyzed (Participants) | 56
  Month 24 | 0.5 (7.11)
  Last Assessment | 0.5 (6.88)

16. Secondary Outcome: Change From Baseline In Hepatic Laboratory Measures For International Normalized Ratio (INR) At Month 6, Month 24, And Last Assessment
Description: The INR was measured over time. Last Assessment was the last available post-baseline result for each participant (ranging from 1 to 24 months).
Time Frame: Baseline through Last Assessment (ranging from 1 to 24 months)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Total
Number analyzed (Participants) | 64
Ratio
  Month 6: number analyzed (Participants) | 56
  Month 6 | -0.02 (0.116)
  Month 24: number analyzed (Participants) | 54
  Month 24 | -0.01 (0.114)
  Last Assessment: number analyzed (Participants) | 62
  Last Assessment | 0.00 (0.114)

17. Secondary Outcome: Change From Baseline In Clinical Global Impression (CGI) Scale Item 1 (Severity Of Illness) At Month 6, Month 24, And Last Assessment
Description: The CGI scale item 1 (severity of illness) rating scale is a commonly used measure of symptom severity, treatment response, and the efficacy of treatments in treatment studies of participants with mental disorders. It uses the Clinical Global Impression - Severity Scale (CGI-S), a 7-point scale that requires the Investigator to rate the severity of the participant's illness at the time of assessment, relative to the Investigator's past experience with participants who had the same diagnosis. Considering total clinical experience, a participant was assessed on severity of illness at the time of rating as: 1, normal, not at all ill; 2, borderline ill; 3, mildly ill; 4, moderately ill; 5, markedly ill; 6, severely ill; or 7, extremely ill. A decrease in score indicates improvement in disease severity. Last Assessment was the last available post-baseline result for each participant (ranging from 1 to 24 months).
Time Frame: Baseline through Last Assessment (ranging from 1 to 24 months)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Total
Number analyzed (Participants) | 64
score on a scale
  Month 6: number analyzed (Participants) | 60
  Month 6 | -0.3 (0.89)
  Month 24: number analyzed (Participants) | 56
  Month 24 | -0.6 (0.97)
  Last Assessment | -0.6 (0.94)

18. Secondary Outcome: CGI Scale Item 2 (Global Improvement) At Month 6, Month 24, And Last Assessment
Description: The CGI scale item 2 (global improvement) is a rating scale commonly used measure of symptom severity, treatment response, and the efficacy of treatments in treatment studies of participants with mental disorders. It uses the Clinical Global Impression - Improvement Scale (CGI-I), a 7-point scale that requires the Investigator to assess how much the participant's illness has improved or worsened relative to the Baseline state at the beginning of the study and rate as: 1, very much improved; 2, much improved; 3, minimally improved; 4, no change; 5, minimally worse; 6, much worse; or 7, very much worse. A decrease in score indicates improvement in disease severity. Last Assessment was the last available post-baseline result for each participant (ranging from 1 to 24 months).
Time Frame: Baseline through Last Assessment (ranging from 1 to 24 months)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Total
Number analyzed (Participants) | 64
score on a scale
  Month 6: number analyzed (Participants) | 60
  Month 6 | 3.3 (1.08)
  Month 24: number analyzed (Participants) | 56
  Month 24 | 3.3 (1.01)
  Last Assessment | 3.4 (0.98)

ADVERSE EVENTS:
Time Frame: From baseline up to 30 months.
Description: Only adverse events (AEs) associated with study-related interventional testing or assessments were collected and summarized by onset, duration, intensity, seriousness, and outcome. AEs not collected included AEs that might have been associated with the specimen collection procedure but resulted only in local, mild or transient discomforts, redness, slight discomfort and AEs related to WD or treatment, or any other medical condition or events experienced during the study, including death.
Arm/Group | Total
All-Cause Mortality (participants affected / at risk) | 1/64
Serious Adverse Events (participants affected / at risk) | 0/64
Other Adverse Events (participants affected / at risk) | 1/64
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Total (N=64)
Haematoma (Vascular disorders) | 1

LIMITATIONS AND CAVEATS:
Only AEs associated with study-related interventional testing or assessments (that is, venipuncture) were collected.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-09-21): https://cdn.clinicaltrials.gov/large-docs/15/NCT02763215/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-17): https://cdn.clinicaltrials.gov/large-docs/15/NCT02763215/SAP_001.pdf